CLINICAL TRIAL: NCT01330147
Title: HPV Prevalence in the Mouth and Oropharynx of the Tonsillectomy Population
Acronym: Oromouth
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: RG12-208; 12344 (Other: NIHR)
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Chronic Tonsillitis
Keywords: HPV; oral cancer; oropharyngeal cancer; tonsillectomy
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral rinse, Oral Mucosal Trasudate, Urine, Whole Blood, Nail brushings, Mouth brush biopsies (scrapes) and Tonsillectomy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tonsillectomy: Subjects undergoing tonsillectomy for non-cancer reasons including operations for: recurrent tonsillitis, asymmetric tonsils, snoring surgery or obstructive sleep apnoea.

SUMMARY:
The principal aim of this study is to provide vital current data on the prevalence, distribution and natural history of Human Papilloma Virus (HPV) infection in the mouth. This data is an essential requirement for the assessment, development and evaluation of cost effectiveness of prophylactic vaccination and screening programmes.

DETAILED DESCRIPTION:
Patients undergoing a tonsillectomy operation for non-cancerous reasons will be recruited for this study. They will be asked to complete two questionnaires (study and sexual practices), provide saliva, urine and a blood sample. Following anaesthesia, oropharyngeal brushings and a tonsillectomy will be performed and all the samples will be processed for evidence of HPV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing tonsillectomy for non cancer reasons including operations for: recurrent tonsillitis, asymmetric tonsils, snoring surgery or obstructive sleep apnoea
2. Age - 0 to 65 years
3. Subject or legal guardian has given informed written consent

Exclusion Criteria:

1. Subjects undergoing adenoidectomy alone with no tonsillectomy
2. Subjects with previous oropharyngeal cancer or oral cancer, or any other head and neck cancer such as nasopharyngeal or laryngeal cancer that is currently undergoing or has previously been diagnosed or treated
3. Learning disability preventing an adult over 16 years old from giving their own consent

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing a tonsillectomy operation for non-cancerous reasons at the hospital will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 937 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of HPV in tonsils and in oral scrape sample | 36 months
  Presence of HPV result

SECONDARY OUTCOMES:
HPV vaccination status | 36 months
  vaccination received yes/no and the type of vaccination description

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, Prof, Principal Investigator — The University of Birmingham
Locations (8):
- United Kingdom (8):
  - University Hospitals Coventry & Warwickshire Trust, Coventry, England
  - University Hospital Birmingham, Birmingham, West Midlands
  - Birmingham City Hospital, Birmingham
  - Birmingham Children Hospital, Birmingham
  - Heartlands Hospital, Birmingham
  - Kidderminster Hospital, Kidderminster
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Undecided